CLINICAL TRIAL: NCT04072887
Title: A 24-week Multi-center, Double-blind, Placebo Controlled Dose-range Finding Study to Investigate the Efficacy and Safety of Oral QBW251 in COPD Patients on Triple Inhaled Therapy (LABA / LAMA / ICS)
Brief Title: Dose-range Finding Efficacy and Safety Study for QBW251 in COPD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQBW251B2201; 2018-003197-28 (EudraCT Number)
Record Dates: First submitted 2019-08-07; First posted 2019-08-28 (Actual); Results first posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — icenticaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- QBW251 450 mg (Experimental): QBW251 was orally administered 450 mg b.i.d for 24 weeks
  Interventions: Drug: QBW251; Drug: COPD maintenance background therapy
- QBW251 300 mg (Experimental): QBW251 was orally administered 300 mg b.i.d for 24 weeks
  Interventions: Drug: QBW251; Drug: COPD maintenance background therapy
- QBW251 150 mg (Experimental): QBW251 was orally administered 150 mg b.i.d for 24 weeks
  Interventions: Drug: QBW251; Drug: COPD maintenance background therapy
- QBW251 75 mg (Experimental): QBW251 was orally administered 75 mg b.i.d for 24 weeks
  Interventions: Drug: QBW251; Drug: COPD maintenance background therapy
- QBW251 25 mg (Experimental): QBW251 was orally administered 25 mg b.i.d for 24 weeks
  Interventions: Drug: QBW251; Drug: COPD maintenance background therapy
- Placebo (Placebo Comparator): Placebo was orally administered b.i.d for 24 weeks
  Interventions: Drug: Placebo; Drug: COPD maintenance background therapy

INTERVENTIONS:
Drug: QBW251 — QBW251 oral capsules (450, 300, 150, 75 and 25 mg) of identical appearance to ensure blinding administered twice a day (b.i.d) for 24 weeks
  Arms: QBW251 150 mg; QBW251 25 mg; QBW251 300 mg; QBW251 450 mg; QBW251 75 mg
Drug: Placebo — Placebo oral capsules administered twice a day for 24 weeks
  Arms: Placebo
Drug: COPD maintenance background therapy — Combination of fluticasone furoate, vilanterol and umeclidinium bromide

SUMMARY:
This clinical study was designed to support the dose selection for future studies by evaluating efficacy and safety of different QBW251 doses in Chronic obstructive pulmonary disease (COPD) patients with chronic bronchitis and a history of exacerbations, compared to placebo, when added to a triple inhaled therapy of LABA, LAMA and ICS.

DETAILED DESCRIPTION:
This study used a 6 treatment arm, parallel-group, randomized, double-blind study design. 974 male and female COPD patients were randomized into the trial. The study consisted of four distinct study periods:

* Screening (Weeks -3 to -2): Participants underwent a screening period of 1 week where were assessed for eligibility and tapered off disallowed medications.
* Run-in (Days -14 to 1): Subsequently, participants entered the run-in period of up to 2 weeks to establish baseline values for symptom assessments, to standardize the COPD background therapy (triple combination LABA/LAMA/ICS), and to complete eligibility assessments.
* Treatment (Day 1 to Week 24): Eligible participants moved into the Day 1 visit where they were stratified according to their smoking status (current or ex-smoker) and severity of airflow limitation (FEV1 ≥ 30% to < 50% and ≥ 50% to < 80%) and then randomized into 1 of 6 treatment arms with a randomization ratio of 2:2:1:1:1:2 (450 mg b.i.d., 300 mg b.i.d., 150 mg b.i.d., 75 mg b.i.d., 25 mg b.i.d., placebo). The treatment period consisted of 24 weeks, during which the participant returned to the site for regular visits (Day 1 - Week 24). QBW251 450 mg arm was discontinued early based on a pre-defined pharmacokinetic exposure stopping rule.
* Follow-up (Weeks 25-28): Upon completion of the treatment period, participants were followed up for safety assessments for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female COPD patients aged ≥40 years, who have signed an Informed Consent Form prior to initiation of any study-related procedure.
* Current or ex-smokers who have a smoking history of at least 10 pack years.
* Patients who have been treated with a triple combination of LABA/LAMA/ICS for the last 3 months prior to screening.
* Patients featuring chronic bronchitis

Exclusion Criteria:

* Patients who have had a COPD exacerbation that required treatment with antibiotics and/or oral corticosteroids and/or hospitalization, or a respiratory tract infection in the 4 weeks prior to screening, or between screening and randomization.
* Patients with any documented history of asthma, or with an onset of chronic respiratory symptoms, including a COPD diagnosis, prior to age 40 years.
* Patients with a body mass index (BMI) of more than 40 kg/m2.
* Use of other investigational drugs (approved or unapproved) within 30 days or 5 half-lives prior to screening, or until the expected pharmacodynamic effect has returned to baseline (e.g., biologics), whichever is longer; or longer if required by local regulations.
* Pregnant or nursing (lactating) women, and women of childbearing potential not willing to use acceptable effective methods of contraception during study participation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 974 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (137):
- United States (25):
  - Novartis Investigative Site, Andalusia, Alabama
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Westminster, California
  - Novartis Investigative Site, Ormond Beach, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Florence, Kentucky
  - Novartis Investigative Site, Crowley, Louisiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Zachary, Louisiana
  - Novartis Investigative Site, Livonia, Michigan
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Gastonia, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, McKinney, Texas
  - Novartis Investigative Site, Midlothian, Virginia
- Argentina (8):
  - Novartis Investigative Site, Berazategui, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Concepción del Uruguay, Entre Ríos Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Ciudad Autonoma de Bs As
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Salta
  - Novartis Investigative Site, Santa Fe
- Australia (4):
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Footscray, Victoria
  - Novartis Investigative Site, Spearwood, Western Australia
- Austria (3):
  - Novartis Investigative Site, Feldbach
  - Novartis Investigative Site, Grieskirchen
  - Novartis Investigative Site, Thalheim bei Wels
- Belgium (3):
  - Novartis Investigative Site, Erpent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Canada (3):
  - Novartis Investigative Site, Sherwood Park, Alberta
  - Novartis Investigative Site, Saint-Charles-Borromée, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Novartis Investigative Site, Zipaquirá, Cundinamarca, Colombia
- Czechia (4):
  - Novartis Investigative Site, Liberec, Czech Republic
  - Novartis Investigative Site, Ostrava Poruba, Czech Republic
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Varnsdorf
- Denmark (3):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Hvidovre
- France (4):
  - Novartis Investigative Site, Montpellier, Herault
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Reims
- Germany (10):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Landsberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Mittweida
  - Novartis Investigative Site, Witten
- Greece (2):
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Thessaloniki, GR
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City, GTM
  - Novartis Investigative Site, Guatemala City
- Hong Kong (2):
  - Novartis Investigative Site, New Territories, Hong Kong
  - Novartis Investigative Site, Pokfulam, Hong Kong
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigative Site, Komárom
  - Novartis Investigative Site, Makó
  - Novartis Investigative Site, Pécs
- Italy (3):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Negrar, VR
- Japan (26):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kasuga, Fukuoka
  - Novartis Investigative Site, Koga, Fukuoka
  - Novartis Investigative Site, Yanagawa, Fukuoka
  - Novartis Investigative Site, Mizunami, Gifu
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Naka-gun, Ibaraki
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Matsusaka, Mie-ken
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kawachi-Nagano, Osaka
  - Novartis Investigative Site, Kishiwada, Osaka
  - Novartis Investigative Site, Toyonaka, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Setagaya-Ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shinagawa, Tokyo
  - Novartis Investigative Site, Toshima Ku, Tokyo
  - Novartis Investigative Site, Yamagata, Yamagata
  - Novartis Investigative Site, Osaka
- Netherlands (2):
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Harderwijk
- Philippines (5):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Iloilo City, Iloilo
  - Novartis Investigative Site, Bulacan
  - Novartis Investigative Site, Iloilo City
  - Novartis Investigative Site, Manila
- Poland (3):
  - Novartis Investigative Site, Grudziądz
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Zawadzkie
- Slovakia (7):
  - Novartis Investigative Site, Bardejov, Slovak Republic
  - Novartis Investigative Site, Bojnice, Slovak Republic
  - Novartis Investigative Site, Humenné, Slovak Republic
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Spišská Nová Ves
  - Novartis Investigative Site, Vyšné Hágy
- South Korea (3):
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Incheon
- Spain (3):
  - Novartis Investigative Site, Marbella, Andalusia
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Girona
- Thailand (3):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Mersin
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Martinez FJ, Criner GJ, Gessner C, Jandl M, Scherbovsky F, Shinkai M, Siler TM, Vogelmeier CF, Voves R, Wedzicha JA, Bartels C, Bottoli I, Byiers S, Cardenas P, Eckert JH, Gutzwiller FS, Knorr B, Kothari M, Parlikar R, Tanase AM, Franssen FME. Icenticaftor, a CFTR Potentiator, in COPD: A Multicenter, Parallel-Group, Double-Blind Clinical Trial. Am J Respir Crit Care Med. 2023 Aug 15;208(4):417-427. doi: 10.1164/rccm.202303-0458OC. PMID 37411039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 149 sites in 26 countries.
Pre-assignment Details: Participants underwent a Screening period of up to 1 week. Then, participants entered the run-in period of up to 2 weeks to establish baseline values for symptom assessments, to standardize the COPD background therapy and to complete eligibility assessments.
Period: Overall Study
Arm/Group | QBW251 450 mg | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg | Placebo
Started (All randomized participants) | 99 | 250 | 124 | 126 | 124 | 251
Pharmacokinetic (PK) Set (All randomized participants who have at least one evaluable concentration data sample) | 99 | 250 | 123 | 126 | 124 | 0
Serial Pharmacokinetic (PK) Set (The Serial PK set includes the participants who consented to participate in the PK serial subgroup) | 14 | 21 | 14 | 13 | 14 | 0
Completed | 91 (QBW251 450 mg arm was discontinued early based on a pre-defined pharmacokinetic exposure stopping rule.) | 233 | 122 | 117 | 118 | 236
Not Completed | 8 | 17 | 2 | 9 | 6 | 15
Not completed — Withdrawal by Subject | 3 | 8 | 1 | 3 | 3 | 13
Not completed — Adverse Event | 2 | 4 | 1 | 4 | 0 | 1
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 2 | 0 | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QBW251 450 mg | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg | Placebo | Total
Number analyzed (Participants) | 99 | 250 | 124 | 126 | 124 | 251 | 974
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (7.28) | 66.6 (7.56) | 66.7 (6.58) | 65.7 (8.30) | 67.0 (7.83) | 66.7 (7.59) | 66.6 (7.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 99 | 47 | 50 | 49 | 92 | 373
  Male | 63 | 151 | 77 | 76 | 75 | 159 | 601
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 10 | 1 | 4 | 4 | 5 | 26
  Asian | 9 | 42 | 27 | 20 | 25 | 43 | 166
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 2 | 6 | 2 | 5 | 21
  White | 87 | 193 | 94 | 96 | 93 | 198 | 761
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) at Week 12
Description: The primary efficacy analysis assessed the effect of QBW251 on the absolute change from baseline in trough FEV1 in liters on Week 12. Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Baseline measurement was defined as the baseline visit pre-bronchodilator spirometry assessment.
  Change from baseline in the FEV1 mean scores were analyzed using a Mixed Model for Repeated Measures (MMRM): treatment + baseline score + smoking status at screening + run-in FEV1 + airflow limitation severity + region + time interval + treatment*time interval interaction + baseline score*time interval interaction.
Time Frame: Baseline and Week 12
Population: The overall number of participants analyzed includes all randomized participants with a value at both baseline and week 12. Results for the QBW251 450 mg arm need to be interpreted with caution as the arm was discontinued early based on a pre-defined pharmacokinetic exposure stopping rule.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | QBW251 450 mg | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg | Placebo
Number analyzed (Participants) | 42 | 209 | 111 | 112 | 105 | 219
Liter | 0.013 (0.021) | 0.013 (0.0103) | 0.014 (0.0142) | 0.021 (0.0141) | 0.006 (0.0144) | 0.001 (0.0101)
Statistical Analysis 1: Comparison: QBW251 450 mg vs Placebo; Test type: Superiority; p = 0.628, ANCOVA; Least Squares Mean Difference = 0.011, 90% CI 2-sided [-0.027 to 0.050], Standard Error of Mean 0.0235
Statistical Analysis 2: Comparison: QBW251 300 mg vs Placebo; Test type: Superiority; p = 0.425, ANCOVA; Least Squares Mean Difference = 0.012, 90% CI 2-sided [-0.012 to 0.035], Standard Error of Mean 0.0144
Statistical Analysis 3: Comparison: QBW251 150 mg vs Placebo; Test type: Superiority; p = 0.463, ANCOVA; Least Squares Mean Difference = 0.013, 90% CI 2-sided [-0.016 to 0.041], Standard Error of Mean 0.0174
Statistical Analysis 4: Comparison: QBW251 75 mg vs Placebo; Test type: Superiority; p = 0.244, ANCOVA; Least Squares Mean Difference = 0.020, 90% CI 2-sided [-0.008 to 0.049], Standard Error of Mean 0.0173
Statistical Analysis 5: Comparison: QBW251 25 mg vs Placebo; Test type: Superiority; p = 0.793, ANCOVA; Least Squares Mean Difference = 0.005, 90% CI 2-sided [-0.024 to 0.034], Standard Error of Mean 0.0176

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1)
Description: The primary efficacy analysis assessed the effect of QBW251 on the absolute change from baseline in trough FEV1 in liters compared to placebo on Weeks 4, 8, 16, 20 and 24. Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Baseline measurement was defined as the baseline visit pre-bronchodilator spirometry assessment. A positive trend for change from baseline in FEV1 across the dose range is considered a favorable outcome.
Time Frame: Baseline, weeks 4, 8, 16, 20 and 24
Population: The overall number of participants analyzed includes all randomized participants. The number analyzed per row represents participants with evaluable data at each time point. Results for the QBW251 450 mg arm need to be interpreted with caution as the arm was discontinued early based on a pre-defined pharmacokinetic exposure stopping rule.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | QBW251 450 mg | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg | Placebo
Number analyzed (Participants) | 80 | 224 | 115 | 117 | 114 | 221
Liter
  Week 4 | 0.007 (0.14) | 0.007 (0.15) | 0.009 (0.13) | 0.000 (0.14) | 0.009 (0.14) | 0.005 (0.13)
  Week 8: number analyzed (Participants) | 61 | 216 | 110 | 113 | 111 | 221
  Week 8 | 0.028 (0.14) | 0.013 (0.16) | -0.002 (0.13) | 0.002 (0.15) | 0.016 (0.16) | 0.009 (0.15)
  Week 16: number analyzed (Participants) | 32 | 209 | 107 | 109 | 104 | 214
  Week 16 | 0.013 (0.18) | 0.003 (0.16) | 0.005 (0.14) | 0.011 (0.15) | 0.007 (0.17) | -0.011 (0.14)
  Week 20: number analyzed (Participants) | 23 | 199 | 105 | 108 | 102 | 211
  Week 20 | -0.031 (0.20) | 0.005 (0.18) | 0.012 (0.13) | 0.001 (0.16) | 0.003 (0.16) | -0.007 (0.15)
  Week 24: number analyzed (Participants) | 11 | 195 | 109 | 106 | 98 | 212
  Week 24 | 0.033 (0.13) | 0.023 (0.19) | 0.004 (0.16) | 0.003 (0.19) | 0.003 (0.17) | -0.013 (0.16)

3. Secondary Outcome: Change From Baseline in Evaluating Respiratory Symptoms (E-RS); Total Score
Description: The E-RS assesses overall daily respiratory COPD symptoms (Total score) and it is derived as the sum of 11 severity items; a higher scores indicate more severe symptoms. E-RS total score has a range of 0 to 40.
  Change from baseline in the E-RS Total weekly mean scores were analyzed using a Mixed Model for Repeated Measures (MMRM): treatment + baseline score + smoking status at screening + run-in E-RS + airflow limitation severity + region + time interval + treatment*time interval interaction + baseline score*time interval interaction.
  The mean baseline E-RS Total score was the average of the corresponding daily scores from the run-in period.
  A negative change from baseline corresponds to improvement in symptoms severity.
Time Frame: Baseline, weeks 12 and 24
Population: The overall number of participants analyzed includes all randomized participants. The number analyzed per row represents participants with evaluable data at each time point. QBW251 450 mg arm was excluded from the analysis as it was discontinued early based on a pre-defined pharmacokinetic exposure stopping rule.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg | Placebo
Number analyzed (Participants) | 196 | 106 | 112 | 105 | 214
Score on a scale
  Week 12 | -1.75 (0.234) | -1.26 (0.323) | -1.66 (0.317) | -1.30 (0.324) | -1.41 (0.228)
  Week 24: number analyzed (Participants) | 175 | 99 | 98 | 92 | 193
  Week 24 | -2.16 (0.239) | -1.37 (0.327) | -1.36 (0.325) | -1.36 (0.333) | -1.31 (0.232)

4. Secondary Outcome: Change From Baseline in Evaluating Respiratory Symptoms (E-RS); Cough and Sputum Score
Description: The E-RS assesses both overall daily respiratory COPD symptoms (Total score) and specific respiratory symptoms using 3 subscales (Breathlessness, Cough & Sputum, and Chest Symptoms). The E-RS comprises 11 severity items and higher scores indicate more severe symptoms. The Cough and Sputum subscale score has a range of 0 to 11 and was derived as the sum of items 2 - 4.
  Change from baseline in the E-RS Cough and Sputum weekly mean scores were analyzed using a Mixed Model for Repeated Measures (MMRM): treatment + baseline score + smoking status at screening + run-in E-RS + airflow limitation severity + region + time interval + treatment*time interval interaction + baseline score*time interval interaction.
  The mean baseline E-RS Cough & Sputum subscale score was the average of the corresponding daily scores from the run-in period. Lower scores in the change from baseline correspond to lower symptom severity.
Time Frame: Baseline, weeks 12 and 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg | Placebo
Number analyzed (Participants) | 196 | 106 | 112 | 105 | 214
Score on a scale
  Week 12 | -0.78 (0.077) | -0.63 (0.105) | -0.52 (0.104) | -0.22 (0.106) | -0.44 (0.074)
  Week 24: number analyzed (Participants) | 175 | 99 | 98 | 92 | 193
  Week 24 | -0.90 (0.078) | -0.68 (0.107) | -0.51 (0.106) | -0.26 (0.109) | -0.50 (0.076)

5. Secondary Outcome: Number of Participants With a "Better" Change in the Patient Global Impression of Severity (PGI-S) From Baseline
Description: The PGI-S questionnaire is a patient-reported outcomes score that rates the severity of the respiratory symptoms and of cough and mucus. The change in severity scores (Better, No change and Worse) from baseline were reported at weeks 12 and 24. Thus, the number of participants with a Better change in the severity score are reported in the table below.
Time Frame: Baseline, weeks 12 and 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg | Placebo
Number analyzed (Participants) | 218 | 116 | 114 | 108 | 218
Participants
  Week 12 - Respiratory Symptoms | 66 | 27 | 35 | 33 | 64
  Week 24 - Respiratory Symptoms: number analyzed (Participants) | 204 | 113 | 109 | 102 | 216
  Week 24 - Respiratory Symptoms | 72 | 28 | 40 | 31 | 79
  Week 12 - Cough and mucus | 85 | 55 | 54 | 41 | 78
  Week 24 - Cough and mucus | 104 | 57 | 50 | 37 | 96

6. Secondary Outcome: Change From Baseline in the Cough and Sputum Assessment Questionnaire (CASA-Q)
Description: The CASA-Q is a validated questionnaire instrument used to measure cough and sputum production, and their impact in patients COPD and/or chronic bronchitis. It contains a total of 20 items on a 5-step scale distributed in 4 domains: Cough symptoms, Cough impact, Sputum symptoms and Sputum impact. All items are rescored from 1-5 to 0-4 and then reverse scored such that better responses have higher scores. The four domains are ranged from 0-100 where higher scores associated with fewer symptoms/less impact due to cough or sputum.
  Change from baseline in the CASA-Q cough and symptoms scores were analyzed using a Mixed Model for Repeated Measures (MMRM): treatment + baseline score + smoking status at screening + run-in E-RS + airflow limitation severity + region + time interval + treatment*time interval interaction + baseline score*time interval interaction.
Time Frame: Baseline, weeks 12 and 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg | Placebo
Number analyzed (Participants) | 217 | 115 | 114 | 108 | 218
Score on a scale
  Cough symptoms score, week 12 | 6.06 (1.082) | 8.82 (1.488) | 6.68 (1.498) | 6.73 (1.535) | 6.06 (1.077)
  Cough symptoms score, week 24: number analyzed (Participants) | 204 | 112 | 109 | 102 | 216
  Cough symptoms score, week 24 | 10.49 (1.148) | 10.59 (1.556) | 8.04 (1.575) | 5.84 (1.623) | 7.25 (1.118)
  Cough impact score, week 12 | 4.97 (0.983) | 5.94 (1.352) | 5.89 (1.359) | 5.03 (1.394) | 5.26 (0.978)
  Cough impact score, week 24: number analyzed (Participants) | 204 | 112 | 109 | 102 | 216
  Cough impact score, week 24 | 7.08 (0.983) | 8.29 (1.334) | 7.51 (1.349) | 4.02 (1.391) | 7.12 (0.958)
  Sputum symptoms score, week 12 | 7.74 (1.142) | 8.51 (1.571) | 7.01 (1.580) | 5.74 (1.620) | 6.96 (1.136)
  Sputum symptoms score, week 24: number analyzed (Participants) | 204 | 112 | 109 | 102 | 216
  Sputum symptoms score, week 24 | 10.52 (1.242) | 11.34 (1.685) | 5.81 (1.704) | 4.64 (1.756) | 9.05 (1.211)
  Sputum impact score, week 12 | 5.88 (1.011) | 6.58 (1.391) | 6.98 (1.398) | 4.35 (1.433) | 4.72 (1.005)
  Sputum impact score, week 24: number analyzed (Participants) | 204 | 112 | 109 | 102 | 216
  Sputum impact score, week 24 | 7.14 (1.032) | 7.66 (1.401) | 7.75 (1.417) | 4.40 (1.460) | 7.04 (1.007)

7. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire (SGRQ)
Description: SGRQ measures health impairment and contains 50 items divided into three components: Symptoms, Activity and Impacts. A score was calculated for each component and a "Total" score was also calculated. In each case the lowest possible value is zero and the highest 100. Higher values correspond to greater impairment of quality of life.
  Change from baseline in the SGRQ scores were analyzed using a Mixed Model for Repeated Measures (MMRM): treatment + baseline score + smoking status at screening + baseline SGRQ score + airflow limitation severity + region + time interval + treatment*time interval interaction + baseline score*time interval interaction.
Time Frame: Baseline, weeks 12 and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QBW251 450 mg | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg | Placebo
Number analyzed (Participants) | 48 | 222 | 117 | 116 | 111 | 221
Score on a scale
  Week 12 - Total score | -0.34 (11.17) | -5.84 (14.82) | -3.14 (12.67) | -6.78 (14.64) | -3.85 (10.82) | -3.36 (13.27)
  Week 24 - Total score: number analyzed (Participants) | 12 | 206 | 114 | 110 | 104 | 219
  Week 24 - Total score | -2.93 (10.58) | -6.48 (15.35) | -3.69 (12.39) | -6.06 (14.88) | -1.70 (10.97) | -4.37 (13.00)
  Week 12 - Symptoms score | -5.24 (21.16) | -8.23 (18.73) | -5.70 (18.39) | -6.93 (19.29) | -5.59 (16.52) | -6.07 (17.14)
  Week 24 - Symptoms score: number analyzed (Participants) | 12 | 206 | 114 | 110 | 104 | 219
  Week 24 - Symptoms score | -7.90 (22.47) | -10.59 (21.06) | -7.09 (17.02) | -8.42 (18.21) | -5.16 (15.61) | -6.97 (17.39)
  Week 12 - Activity score | -2.00 (10.83) | -4.80 (17.67) | -4.72 (17.35) | -7.27 (17.48) | -4.06 (14.68) | -2.40 (15.21)
  Week 24 - Activity score: number analyzed (Participants) | 12 | 206 | 114 | 110 | 104 | 219
  Week 24 - Activity score | -1.25 (12.50) | -5.12 (17.36) | -3.69 (16.37) | -5.80 (20.47) | -1.20 (14.36) | -4.27 (16.07)
  Week 12 - Impacts score | 2.03 (14.28) | -5.69 (17.06) | -1.49 (13.88) | -6.42 (16.63) | -3.13 (13.11) | -3.11 (15.90)
  Week 24 - Impacts score: number analyzed (Participants) | 12 | 206 | 114 | 110 | 104 | 219
  Week 24 - Impacts score | -2.21 (8.24) | -6.04 (17.455) | -2.63 (14.18) | -5.44 (16.05) | -1.04 (13.95) | -3.68 (14.95)

8. Secondary Outcome: Minimum Plasma Concentration (Cmin) for QBW251
Description: Venous whole blood samples were collected for pharmacokinetics characterization. Cmin was measured pre dose at all visits and was summarized using descriptive statistics. All concentrations below the lower limit of quantification (LLOQ) were treated as zero.
Time Frame: Pre-dose on Days 15, 29, 57, 85, 113, 141 and 169
Population: The overall number of participants analyzed includes the PK analysis set. The number analyzed per row represents participants with evaluable data at each time point. Results for the QBW251 450 mg arm need to be interpreted with caution as the arm was discontinued early based on a pre-defined pharmacokinetic exposure stopping rule.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBW251 450 mg | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg
Number analyzed (Participants) | 75 | 180 | 101 | 100 | 96
ng/mL
  Day 15 | 1280 (1700) | 619 (1230) | 143 (158) | 44.0 (49.0) | 12.7 (15.5)
  Day 29: number analyzed (Participants) | 61 | 179 | 96 | 91 | 83
  Day 29 | 951 (1050) | 571 (923) | 125 (123) | 47.8 (47.3) | 10.1 (10.1)
  Day 57: number analyzed (Participants) | 53 | 163 | 89 | 90 | 86
  Day 57 | 1040 (1330) | 572 (833) | 116 (103) | 47.7 (62.2) | 14.2 (25.5)
  Day 85: number analyzed (Participants) | 37 | 165 | 85 | 81 | 74
  Day 85 | 1080 (1360) | 587 (951) | 119 (147) | 49.7 (71.2) | 9.93 (10.3)
  Day 113: number analyzed (Participants) | 27 | 161 | 90 | 87 | 85
  Day 113 | 859 (1150) | 593 (1000) | 120 (130) | 52.7 (73.9) | 9.89 (9.20)
  Day 141: number analyzed (Participants) | 22 | 167 | 92 | 91 | 85
  Day 141 | 1150 (1150) | 552 (923) | 118 (103) | 66.8 (226) | 15.9 (45.7)
  Day 169: number analyzed (Participants) | 5 | 167 | 95 | 82 | 84
  Day 169 | 637 (349) | 465 (618) | 128 (147) | 44.9 (61.1) | 8.97 (8.08)

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) for QBW251
Description: Venous whole blood samples were collected for pharmacokinetics characterization. Cmax was calculated from plasma concentration data using non-compartmental methods and summarized using descriptive statistics. Cmax was measured in the samples taken at 3 hours post-dose with the exception of the participants included in the Serial PK set on Days 1 and 15 for whom all samples (1, 2, 4, 6, and 8 hours post-dose) were taken into consideration for the measurement of Cmax. All concentrations below the lower limit of quantification (LLOQ) were treated as zero.
Time Frame: Days 1, 15 and 169
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBW251 450 mg | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg
Number analyzed (Participants) | 93 | 222 | 110 | 115 | 124
ng/mL
  Day 1 | 1280 (847) | 751 (598) | 251 (238) | 68.9 (64.5) | 14.4 (15.2)
  Day 15: number analyzed (Participants) | 75 | 198 | 107 | 111 | 108
  Day 15 | 2500 (1710) | 1320 (1030) | 411 (368) | 114 (101) | 26.1 (20.6)
  Day 169: number analyzed (Participants) | 6 | 182 | 102 | 88 | 98
  Day 169 | 2370 (1160) | 1210 (797) | 361 (303) | 104 (86.6) | 22.5 (16.4)

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) for QBW251 in Serial PK Set
Description: Venous whole blood samples were collected for pharmacokinetics characterization. Cmax was calculated from plasma concentration data using non-compartmental methods and summarized using descriptive statistics. All concentrations below the lower limit of quantification (LLOQ) were treated as zero.
Time Frame: 1, 2, 4, 6, and 8 hours post-dose on Days 1 and 15
Population: The overall number of participants analyzed includes the Serial PK analysis set. The number analyzed per row represents participants with evaluable data at each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBW251 450 mg | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg
Number analyzed (Participants) | 14 | 16 | 13 | 13 | 13
ng/mL
  Day 1 | 1510 (928) | 1280 (622) | 478 (241) | 96.6 (72.7) | 25.3 (29.7)
  Day 15: number analyzed (Participants) | 12 | 15 | 13 | 13 | 13
  Day 15 | 2700 (1170) | 1870 (844) | 542 (523) | 175 (127) | 39.4 (27.0)

11. Secondary Outcome: Area Under the Curve From Time 0 to 24 Hours (AUC0-24h) of QBW251 in Serial PK Set
Description: Venous whole blood samples were collected for pharmacokinetics characterization. AUC0-24h was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics. All concentrations below the lower limit of quantification (LLOQ) were treated as zero.
Time Frame: 1, 2, 4, 6, and 8 hours post-dose on Days 1 and 15
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | QBW251 450 mg | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg
Number analyzed (Participants) | 11 | 14 | 11 | 12 | 12
ng*h/mL
  Day 1: number analyzed (Participants) | 11 | 14 | 11 | 9 | 9
  Day 1 | 10900 (3740) | 8480 (3660) | 2920 (1140) | 769 (330) | 185 (107)
  Day 15: number analyzed (Participants) | 10 | 14 | 10 | 12 | 12
  Day 15 | 30000 (22600) | 16500 (8380) | 4740 (2390) | 1390 (679) | 333 (209)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the start of treatment to 30 days after end of treatment, assessed up to maximum duration of 199 days.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Groups:
- Total: Total
Arm/Group | QBW251 450 mg | QBW251 300 mg | QBW251 150 mg | QBW251 75 mg | QBW251 25 mg | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/99 | 2/250 | 0/124 | 2/126 | 3/124 | 0/251 | 7/974
Serious Adverse Events (participants affected / at risk) | 10/99 | 33/250 | 6/124 | 14/126 | 12/124 | 15/251 | 90/974
Other Adverse Events (participants affected / at risk) | 48/99 | 117/250 | 59/124 | 55/126 | 60/124 | 107/251 | 446/974
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QBW251 450 mg (N=99) | QBW251 300 mg (N=250) | QBW251 150 mg (N=124) | QBW251 75 mg (N=126) | QBW251 25 mg (N=124) | Placebo (N=251) | Total (N=974)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cor pulmonale (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vascular stent thrombosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 3 | 0 | 1 | 2 | 0 | 6
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Peritoneal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 6 | 0 | 3 | 2 | 3 | 15
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bone graft lysis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 0 | 0 | 0 | 4
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Non-small cell lung cancer stage IIIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 9 | 1 | 5 | 2 | 5 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QBW251 450 mg (N=99) | QBW251 300 mg (N=250) | QBW251 150 mg (N=124) | QBW251 75 mg (N=126) | QBW251 25 mg (N=124) | Placebo (N=251) | Total (N=974)
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 2 | 0 | 1 | 3 | 9
Diarrhoea (Gastrointestinal disorders) | 6 | 7 | 1 | 2 | 3 | 6 | 25
Nausea (Gastrointestinal disorders) | 5 | 4 | 2 | 3 | 1 | 5 | 20
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 3 | 1 | 4 | 11
Chest pain (General disorders) | 0 | 2 | 3 | 0 | 1 | 1 | 7
Fatigue (General disorders) | 2 | 3 | 2 | 1 | 0 | 3 | 11
Bronchitis (Infections and infestations) | 4 | 6 | 2 | 0 | 3 | 2 | 17
COVID-19 (Infections and infestations) | 0 | 4 | 1 | 1 | 6 | 5 | 17
Cystitis (Infections and infestations) | 0 | 2 | 2 | 3 | 1 | 1 | 9
Gastroenteritis (Infections and infestations) | 4 | 2 | 0 | 1 | 1 | 1 | 9
Influenza (Infections and infestations) | 2 | 4 | 0 | 1 | 1 | 2 | 10
Lower respiratory tract infection (Infections and infestations) | 3 | 3 | 3 | 2 | 4 | 5 | 20
Nasopharyngitis (Infections and infestations) | 4 | 12 | 5 | 10 | 6 | 10 | 47
Pharyngitis (Infections and infestations) | 2 | 0 | 1 | 0 | 2 | 3 | 8
Pneumonia (Infections and infestations) | 3 | 5 | 1 | 1 | 2 | 2 | 14
Sinusitis (Infections and infestations) | 0 | 1 | 3 | 1 | 0 | 2 | 7
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 5 | 0 | 0 | 5 | 17
Upper respiratory tract infection bacterial (Infections and infestations) | 3 | 12 | 4 | 4 | 4 | 9 | 36
Urinary tract infection (Infections and infestations) | 3 | 8 | 3 | 5 | 2 | 5 | 26
Viral upper respiratory tract infection (Infections and infestations) | 3 | 8 | 3 | 3 | 3 | 7 | 27
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 3 | 1 | 6
C-reactive protein increased (Investigations) | 1 | 8 | 4 | 0 | 0 | 2 | 15
Gamma-glutamyltransferase increased (Investigations) | 4 | 6 | 4 | 2 | 0 | 3 | 19
Haemoglobin decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 1 | 3
Hepatic enzyme increased (Investigations) | 2 | 2 | 0 | 0 | 0 | 2 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 1 | 3 | 6 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7 | 3 | 3 | 2 | 7 | 24
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 1 | 0 | 3 | 10
Dizziness (Nervous system disorders) | 4 | 5 | 0 | 1 | 1 | 1 | 12
Headache (Nervous system disorders) | 4 | 11 | 4 | 4 | 4 | 6 | 33
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 | 51 | 32 | 24 | 34 | 56 | 213
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 1 | 1 | 6 | 13
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 3
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 0 | 0 | 0 | 7
Hypertension (Vascular disorders) | 4 | 8 | 3 | 3 | 3 | 4 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT04072887/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT04072887/SAP_001.pdf